CLINICAL TRIAL: NCT06557551
Title: Prophylactic Surfactant by Thin Endotracheal Catheter for Preterm Infants At Birth: the ProTeCt Trial
Acronym: proTeCt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: proTeCt 01
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Infant, Newborn, Diseases; Prematurity; Prematurity; Extreme; Respiratory Distress Syndrome in Premature Infant
MeSH Terms: conditions — Infant, Newborn, Diseases; Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomised, open-label, parallel group group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thin catheter surfactant (Experimental): At or after 5 minutes of life, participants will have a thin endotracheal catheter (Surfcath, Vygon, Ecouen, France) inserted under video laryngoscopy (C-MAC, Karl Storz, Tuttlingen, Germany), through which they will receive surfactant (Curosurf, Chiesi Farmaceutici, Parma, Italy - 120mg for infants < 26 weeks, 240mg for infants 26 - 27+6 weeks). The catheter will then be removed, and they will continue on face mask breathing support.
  Interventions: Other: Thin catheter surfactant
- Standard care (No Intervention): Participants will continue on face mask breathing support.

INTERVENTIONS:
Other: Thin catheter surfactant — Surfactant given through thin catheter inserted under video laryngoscopy at or after 5 minutes of life
  Arms: Thin catheter surfactant

SUMMARY:
The goal of this clinical trial is to learn whether giving surfactant through a thin endotracheal catheter to extremely premature babies shortly after birth reduces the number of them who are ventilated in the first 3 days of life.

The main question it aims to answer is:

Do fewer babies who receive prophylactic thin catheter surfactant under video laryngoscopy shortly after birth go on to be ventilated within 72 hours of birth?

Extremely premature babies who are receiving breathing support through a face mask will either:

* Receive surfactant through a thin catheter that is inserted into their windpipe (trachea) under video laryngoscopy at or after 5 minutes of life, have the catheter removed immediately, and return to face mask breathing support; or
* Continue on face mask breathing support.

All babies will be closely watched to see whether they are ventilated for breathing support in the first 72 hours of life.

DETAILED DESCRIPTION:
Preterm infants - particularly those born before 28 weeks of gestation - are at risk of developing respiratory distress syndrome (RDS), a condition characterised by structural and functional lung immaturity that leads to progressive respiratory failure. Infants at high risk of or who show early signs of RDS are treated with continuous positive airway pressure (CPAP) in an attempt to prevent respiratory failure. Infants whose RDS worsens despite CPAP are given surfactant. To give surfactant, clinicians use a laryngoscope to view the airway and insert a relatively wide-bore endotracheal tube (ETT) directly into the trachea. When an ETT is used to deliver surfactant, the ETT usually remains in place for a period of mechanical ventilation (MV). Clinicians aim to minimise the duration of ventilation, as even short periods of MV may be harmful to the preterm lung. An alternative approach, sometimes called "less-invasive surfactant application" (LISA), is to give surfactant through a thin endotracheal catheter. These thin catheters (TC) cannot be used for mechanical ventilation and so they are immediately removed after the surfactant has been given.

A Cochrane systematic review found that, compared to giving surfactant through an ETT in the NICU, TC surfactant is associated with reduced risk of death or bronchopulmonary dysplasia (BPD), less intubation in the first 72 hours and reduced incidence of major complications and in-hospital mortality. However, the studies included in the systematic review are heterogenous, few of them enrolled infants born before 28 weeks of gestation and none of them evaluated the effects of giving TC surfactant shortly after birth, before starting CPAP in the NICU. In all of these studies, the clinician inserting the TC viewed the airway directly through the mouth (i.e. performed direct laryngoscopy).

Inserting an ETT in a newborn infant using direct laryngoscopy is challenging. Clinicians use clinical signs detected during positive pressure ventilation (PPV) (e.g. detection of exhaled carbon dioxide, auscultation of breath sounds, condensation in the tube in expiration) to determine whether the ETT has been placed correctly. We recently demonstrated that more first intubation attempts with an ETT in newborn infants are successful when clinicians used a video laryngoscope (VL) to view the airway indirectly compared to direct laryngoscopy. . As PPV cannot be given through a TC, the only way of determining the position of a TC is to see it enter the larynx. Using VL during TC insert attempts allows multiple observers to simultaneously and independently determine whether it is in the correct place.

The earlier that surfactant is given, the more effective it appears to be. It is possible that TC surfactant given "prophylactically" - i.e. very shortly after birth, when there are minimal signs of respiratory distress - under VL guidance may substantially reduce the rate of intubation for respiratory failure. If it does, that holds out the prospect that it may reduce rates of the adverse outcomes associated with ventilation (death or BPD etc.) in preterm infants.

ELIGIBILITY:
Inclusion criteria

* Infants of any sex born before 28 weeks of gestation
* Clinicians plan to provide intensive care
* Consent for their participation provided by parent(s)/guardian(s) before their birth

Exclusion criteria

• Major congenital anomalies (e.g. upper airway anomaly, diaphragmatic hernia, gastroschisis, exomphalos major, intestinal atresias, open neural tube defect, aneuploidy, cardiac lesions other than ASD/PFO/VSD/PDA )

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 164 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants intubated in the first 72 hours of life | First 72 hours of life
  Endotracheal intubation
  1. in the Delivery Room for apnoea or bradycardia despite mask PPV; or
  2. in the Neonatal Intensive Care Unit, for 2 or more of
     * worsening clinical signs respiratory distress
     * oxygen requirement > 30% for >30 mins to keep oxygen saturation (SpO2) >90%
     * pH < 7.2 on 2 blood gases 30 minutes apart
     * PCO2 >9kPa on 2 blood gases 30 minutes apart
     * recurrent mask PPV for apnoea
  Participants reach the primary outcome if they are intubated with an endotracheal tube (ETT) for mechanical ventilation, with an ETT for surfactant and mechanical ventilation, with an ETT for surfactant alone, or with a thin catheter for surfactant alone

SECONDARY OUTCOMES:
Number of participants in whom the thin catheter is seen on video laryngoscopy to be successfully inserted at first attempt (intervention group only) | 30 minutes
  Success at first thin catheter insertion attempt (intervention group only)
Number of participants with bradycardia [heart rate (HR) < 100bpm] in the Delivery Room (DR) | 30 minutes
  Bradycardia (HR < 100bpm) in the DR
Number of participants who receive mask Positive Pressure Ventilation (PPV) in the DR | 30 minutes
  Mask PPV in the DR
Number of participants who undergo endotracheal intubation in the DR | 30 minutes
  Endotracheal intubation in the DR
Number of participants who receive chest compressions in the DR | 30 minutes
  Chest compressions in the DR
Number of participants who receive adrenaline in the DR | 30 minutes
  Adrenaline administration in the DR
Number of participants who receive volume expansion in the DR | 30 minutes
  Volume expansion in the DR
Number of participants who are itubated at any time during hospitalisation | 4 months or before hospital discharge, whichever occurs first
  Intubation at any time during hospitalisation
Number if participants who receive intratracheal surfactant post intervention | 4 months or before hospital discharge, whichever occurs first
  Treatment with intratracheal surfactant, post prophylactic delivery room TC surfactant in the intervention group, or at any time in the control group
Number of participants who have pneumothorax drained with needle aspiration or chest drain insertion | 4 months or before hospital discharge, whichever occurs first
  Pneumothorax drained with needle aspiration or chest drain insertion
Duration of mechanical ventilation (days) | 4 months or before hospital discharge, whichever occurs first
  Duration of mechanical ventilation (days)
Duration of any respiratory support (ventilation, CPAP, HFNC) (days) | 4 months or before hospital discharge, whichever occurs first
  Duration of any respiratory support (ventilation, CPAP, HFNC) (days)
Duration of oxygen therapy (days) | 4 months or before hospital discharge, whichever occurs first
  Duration of oxygen therapy (days)
Number of participants who have bronchopulmonary dysplasia (BPD) among survivors to 36 weeks | 4 months or before hospital discharge, whichever occurs first
  Bronchopulmonary dysplasia (BPD) among survivors to 36 weeks
Number of participants who receive postnatal steroids for BPD | 4 months or before hospital discharge, whichever occurs first
  Treatment with systemic postnatal corticosteroids (e.g. dexamethasone) for respiratory insufficiency
Number of participants with severe intraventricular haemorrhage (IVH) (grade III or IV) on cranial ultrasound | 4 months or before hospital discharge, whichever occurs first
  Severe intraventricular haemorrhage (IVH) (grade III or IV) on cranial ultrasound
Number of participants with cystic periventricular leukomalacia (PVL) on cranial ultrasound | 4 months or before hospital discharge, whichever occurs first
  Cystic periventricular leukomalacia (PVL) on cranial ultrasound
Number of participants with patent ductus arteriosus (PDA) treated medically | 4 months or before hospital discharge, whichever occurs first
  Patent ductus arteriosus (PDA) treated medically
Number of participants with PDA treated with transcatheter closure or surgical ligation | 4 months or before hospital discharge, whichever occurs first
  PDA treated with transcatheter closure or surgical ligation
Number of participants with necrotising enterocolitis (NEC) Bell stage 2 or greater | 4 months or before hospital discharge, whichever occurs first
  Necrotising enterocolitis (NEC) Bell stage 2 or greater
Number of participants with spontaneous intestinal perforation (SIP) | 4 months or before hospital discharge, whichever occurs first
  Spontaneous intestinal perforation (SIP)
Number of participants with retinopathy of prematurity (ROP) stage 3 or greater | 4 months or before hospital discharge, whichever occurs first
  Retinopathy of prematurity (ROP) stage 3 or greater
Number of participants who die before or have BPD at 36 weeks | 4 months or before hospital discharge, whichever occurs first
  Death or BPD at 36 weeks
Duration of hospitalisation (days) | 4 months or before hospital discharge, whichever occurs first
  Duration of hospitalisation (days)
Number of participants who are discharged home in oxygen | 4 months or before hospital discharge, whichever occurs first
  Discharged home receiving supplemental oxygen
Number of participants who die during first hospitalisation | 4 months or before hospital discharge, whichever occurs first
  Death during first hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Colm PF O'Donnell, Principal Investigator — National Maternity Hospital, University College Dublin
Locations (1):
- National Maternity Hospital, Dublin, None Selected, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Participant data may be made available to other researchers on receipt of acceptable written request by principal Investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available 1 year after publication for 2 years
Access Criteria: Participant data may be made available to other researchers on receipt of acceptable written request by principal Investigator

REFERENCES:
- [Background] Abdel-Latif ME, Davis PG, Wheeler KI, De Paoli AG, Dargaville PA. Surfactant therapy via thin catheter in preterm infants with or at risk of respiratory distress syndrome. Cochrane Database Syst Rev. 2021 May 10;5(5):CD011672. doi: 10.1002/14651858.CD011672.pub2. PMID 33970483
- [Background] Geraghty LE, Dunne EA, Ni Chathasaigh CM, Vellinga A, Adams NC, O'Currain EM, McCarthy LK, O'Donnell CPF. Video versus Direct Laryngoscopy for Urgent Intubation of Newborn Infants. N Engl J Med. 2024 May 30;390(20):1885-1894. doi: 10.1056/NEJMoa2402785. Epub 2024 May 5. PMID 38709215
- [Background] Bahadue FL, Soll R. Early versus delayed selective surfactant treatment for neonatal respiratory distress syndrome. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD001456. doi: 10.1002/14651858.CD001456.pub2. PMID 23152207